CLINICAL TRIAL: NCT04978974
Title: Stress, Coping Strategies and Quality of Life Among Patients With Chronic Conditions: Implications of Stress Management Program
Brief Title: Implications of Stress Management Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gujrat (Other)
Responsible Party: Principal Investigator, Hafsa Qurban, Mphil Scholar, Priniciple Investigator, Psychologist, Department of Psychology, University of Gujrat, University of Gujrat
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UOG/ASRB/Psych/3/18631/011
Record Dates: First submitted 2021-06-27; First posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Chronic Conditions, Multiple
Keywords: Diabetes; Hypertension; Chronic Condition; Stress Management Program; Perceived Stress; Coping Strategies
MeSH Terms: conditions — Multiple Chronic Conditions; Diabetes Mellitus; Hypertension; Chronic Disease

STUDY DESIGN:
Intervention Model Description: The patients with chronic conditions which included type 2 diabetes and hypertension were selected through purposive sampling technique
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with type 2 Diabetes mellitus and Hypertension (Experimental): patients with type 2 diabetes mellitus and hypertension were selected by using purposive sampling technique to apply stress management program
  Interventions: Behavioral: Stress Management Program

INTERVENTIONS:
Behavioral: Stress Management Program — Stress management program includes different techniques such as relaxation technique, psycho-education, laughing, emotional freedom technique, referenting, cognitive restructuring, rational emotive imagery, time management, anger management, assertiveness and social support

SUMMARY:
Previous studies indicated that patients with diabetes mellitus and hypertension had higher level of perceived stress, used maladaptive coping strategies and poor health-related quality of life. Therefore, stress management program was applied to reduce their perceived stress, improve their coping strategies, improve their health-related quality of life and psychological health of the patients with type 2 diabetes mellitus and hypertension in current study. The main objectives of the current study were to observe the effects of stress management program on perceived stress, coping strategies and health-related quality of life using pre-experimental research design. Patients with diabetes mellitus type 2 and hypertension were selected through purposive sampling technique to apply the eclectic approach of the stress management program. Total 110 patients with type 2 diabetes and hypertension completed the program from 114 patients who gave inform consent for participation in the first session. Perceived stress scale, WHOQOL and Coping strategies questionnaire were administered at the pre and post-levels of the program. Further, base line of targeted domains variables was also filled from the participants at pre, mid and post-levels to access the efficacy of the program which was formulated according to previous research data by the researcher. The stress Management program consisted of 10 session which were delivered to eight groups (diabetic and Hypertensive) in five weeks. Each session had the duration 90 minutes and two sessions were conducted in one week.

ELIGIBILITY:
Inclusion Criteria:

* patients with type II diabetes or hypertension with at least three months duration of illness
* had not attended any psychological intervention or stress management program earlier

Exclusion Criteria:

* Patients who had any other physical/ mental illnesses along with diabetes or hypertension
* Patients with type I diabetes
* Patients with gestational diabetes or hypertension
* Had diabetes or hypertensive condition from less than three month
* Had co morbidity of diabetes and hypertensive chronic conditions

Ages: 31 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2019-05-03 (Actual); Primary Completion 2020-01-03 (Actual); Study Completion 2020-12-29 (Actual)

PRIMARY OUTCOMES:
Effects of stress management program as assessed using Perceived Stress Scale | 10th session (one month and one week from first assessment)
  Consisted of 10 items, Scoring: 0 to 1, The Higher score shows more stress
Effects of stress management program as assessed using Health-Related Quality of Life | 10th session (one month and one week from first assessment)
  Consisted of 26 items, Scoring: 1 to 5, The higher score shows better HRQOL
Effects of stress management program as assessed using Coping Strategies Questionnaire | 10th session (one month and one week from first assessment)
  Consisted of 62 items, Scoring: 1 to 5, The higher score shows high use of coping strategies

SECONDARY OUTCOMES:
Effects of stress management program as assessed using Baseline | base line were used in 5th (two weeks and 3 days) and 10th session (one month and one week from first assessment)
  20 targeted domains which included information about the illness, information about the causes of illness, information about the treatment of illness, efforts to control the level of illness, application of domestic tips, hopefulness, anxiety, negative thoughts, problems in daily activities, problems in social relationships, anger, appetite problems, sleep problems, concentration problems, body pain, fatigue, absent mind, unhealthy diet, loneliness and restlessness at pre, mid and post levels of stress management program. Rating scale ranges from 0-10 (0 shows there is absence of the target construct while 10 shows the high level of target construct).

CONTACTS AND LOCATIONS:
Locations (1):
- Jhelum Poly Clinic, Jhelum, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Due to data confidentiality from the participants, there is no plan of IPD available

REFERENCES:
- [Background] Alshayban D, Joseph R. Health-related quality of life among patients with type 2 diabetes mellitus in Eastern Province, Saudi Arabia: A cross-sectional study. PLoS One. 2020 Jan 10;15(1):e0227573. doi: 10.1371/journal.pone.0227573. eCollection 2020. PMID 31923232